CLINICAL TRIAL: NCT01916460
Title: Intraluminal Endosonography for Examination of the Structural Changes of the Stomach in Gastroparetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E13052
Record Dates: First submitted 2013-06-23; First posted 2013-08-05 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Idiopathic Gastroparesis; Diabetic Gastroparesis
Keywords: Gastroparesis; Endoscopic ultrasound; Interstitial cell of Cajal
MeSH Terms: conditions — Gastroparesis | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gastroparetic patient 19G (Experimental): Endoscopic Ultrasound Fine Needle Aspiration of the gastric wall prior to surgical placement of gastric neurostimulator with 19-gauge fine core needle used for aspiration
  Interventions: Procedure: Endoscopic Ultrasound Fine Needle Aspiration (EUS-FNA)

INTERVENTIONS:
Procedure: Endoscopic Ultrasound Fine Needle Aspiration (EUS-FNA) — After the subjects meet the criteria for enrollment in the study, gastroparetic patients will undergo linear EUS examination of the stomach wall one day prior to their surgery to obtain single or multiple core biopsies of the stomach body wall using the 19-gauge core biopsy needle under EUS guidance. The pathologist will be in the room to assess the adequacy of the sample after each pass. Once the pathologist deemed that the obtained sample is sufficient, the procedure will be terminated

SUMMARY:
Patients who empty their stomach slowly may have what we call "Slow gastric emptying" or "gastroparesis". These patients can have some changes in the thickness of their stomach wall. In addition, they may have loss of some important nerve cells in their stomach muscles. The loss of these cells can cause slow emptying of the stomach. Obtaining a sample from the stomach wall to examine the loss of these cells can help in diagnosing gastroparesis. Up to now, the only way to obtain a tissue sample from the stomach muscle was to undergo an operation in the surgery suite and be hospitalized for several days after the procedure. Usually, we obtain this sample while these patients are having a surgery for another purpose such as placement of a gastric stimulator (a machine which is inserted in the stomach wall to control the stomach rhythm and thus help the stomach to empty faster). Endoscopic ultrasound is an endoscope (a tube with a source of light and ultrasound installed in the tip of the tube) that can measure how thick the stomach wall is and can provide sample "biopsies" of the stomach wall which can be studied for the loss of these specialized muscles and cells.

We are proposing that samples obtained by the endoscopic ultrasound can be sufficient to diagnose "gastroparesis" and can replace the need for obtaining samples by surgery. Endoscopic ultrasound is an outpatient procedure which is not as invasive as surgery.

DETAILED DESCRIPTION:
EUS Fine Needle Aspiration (FNA) Biopsies of the Muscularis Propria (MP) of the gastric wall in patients with gastroparesis (GP) could replace the routine use of surgical full thickness biopsies (FTB) for assessing loss of Interstitial Cell of Cajal (ICC) and cellular infiltrates in the myenteric plexus. The principal investigator investigated the efficacy and safety of EUS Fine Needle Aspiration biopsies of the Muscularis Propria of the stomach antrum in gastroparesis and compared the tissue to a surgically obtained full thickness biopsies in the same patient.

This was a prospective, nonrandomized, feasibility trial. Patients with gastroparesis who were undergoing gastric neurostimulator placement were enrolled. Patients had a gastric wall measurement by radial EUS in the body and antrum of the stomach followed by linear EUS examination and FNA of the muscularis propria in the antrum by using a 19-gauge core needle. Within 24 hours, a full-thickness biopsy specimen of the antrum was obtained surgically during neurostimulator placement. Endoscopic and surgical specimens were compared for tissue morphology, number of ICCs (c-kit stain) and enteric neurons (S-100 stain), and fibrosis (trichome) for each patient. The correlation coefficient of the ICC count per high-power field was used to compare both specimens. Continuous data were compared by using a t test.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age 18 to 80) with objective evidence of gastroparesis who will undergo surgical placement of gastric pacemaker and full thickness gastric wall biopsy. Objective evidence of gastroparesis include the following:

  1. Documented symptoms of gastroparesis for longer than 6 months.
  2. More than 7 episodes of vomiting per week
  3. Refractoriness or intolerance to antiemetics and prokinetic medications
  4. Delayed gastric emptying of solid meal (>60% gastric retention at 2 hours and >10% at 4 hours postprandial) using a standard 4-hour scintigraphic method

Exclusion Criteria:

* Patients with documented organic or intestinal pseudo-obstruction , primary eating or swallowing disorders, rumination syndrome, psychogenic vomiting, cyclic vomiting syndrome, systemic sclerosis, thyroid and adrenal disease, chemical dependency, cancer, peritoneal dialysis, pregnancy.Also, patients with history of gastric surgery such as partial gastric resection or vagatomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The ability of EUS FNA needle to obtain gastric smooth muscle tissue | During the procedure ( 45 minutes)
  Wither FNA needle can obtain sufficient muscularis propria tissue from the gastric wall to perform histological staining for the interstitial cell of Cajal and smooth muscles markers. The specimen from the FNA needle will be compared to the standard full thickness gastric biopsy which is routinely obtained in our institution during the surgical placement of the gastric stimulator.

SECONDARY OUTCOMES:
Safety of EUS FNA of gastric wall ( wither perforation or tear developed after the procedure) | within 24 hours
  The site of EUS FNA in the stomach wall will be examined surgically for perforations and tear during surgical placement of gastric neurostimulator

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed O Othman, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University HSC at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Othman MO, Davis B, Saroseik I, Torabi A, McCallum RW. EUS-guided FNA biopsy of the muscularis propria of the antrum in patients with gastroparesis is feasible and safe. Gastrointest Endosc. 2016 Feb;83(2):327-33. doi: 10.1016/j.gie.2015.06.056. Epub 2015 Aug 28. PMID 26318833